CLINICAL TRIAL: NCT03552627
Title: Perioperative UtiLisation of SupplEmental Oxygen
Acronym: PULSE Ox
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CRI0358
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia
Keywords: hyperoxia; oxygen; surgery; perioperative
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 80% Oxygen (Active Comparator): Patients will receive 80% oxygen throughout anaesthesia in accordance with current World Health Organisation Recommendations
  Interventions: Drug: Oxygen
- 55% Oxygen (Active Comparator): Patients will receive 55% oxygen throughout anaesthesia in accordance with current UK clinical practice
  Interventions: Drug: Oxygen
- 30% Oxygen (Experimental): Patients will receive 30% oxygen throughout anaesthesia in accordance with this research's hypothesis that lowering intraoperative oxygen concentrations may benefit patients
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Medical Oxygen

SUMMARY:
The World Health Organisation recommends that all patients having a general anaesthetic for surgery should be given 80% oxygen as this might reduce their risk of getting an infection after their operation. However there remains a lot of uncertainty about how much oxygen patients should be given whilst undergoing surgery. In other areas of medicine evidence is slowly emerging to suggest that giving less oxygen may be as safe or even safer than giving high amounts of oxygen (e.g. after a heart attack, patients unnecessarily given oxygen seem to do worse than those given air). The amount of oxygen currently given to patients having surgery varies widely; in a recent study of almost 400 procedures across 29 hospitals, we found values ranged from below 30% to almost 100% oxygen. The aim of this research is to explore if giving less oxygen will generate less strain on parts of the body, particularly the lungs as they are always exposed to all of the oxygen that enters the body. Participants undergoing major elective surgical procedures will be randomised to receive either 80%, 55% or 30% throughout their general anaesthetic and levels of inflammation, oxidative stress and perioperative recovery will all be measured for upto 7 days after surgery.

DETAILED DESCRIPTION:
Over 3 million patients receive oxygen (O2) during general anaesthesia (GA) in the UK annually, and a large number of these also have co-morbid respiratory diseases such as Asthma or COPD. The World Health Organisation (WHO) recently recommended that all surgical patients receive 80% O2 throughout GA and for 6 hours in recovery to reduce Surgical Site Infections (SSIs). However, a recent Cochrane systematic review found no evidence of benefit from this approach and some evidence that harm could be increased (including mortality).

Excess oxygen has been associated with worse outcomes in many areas of medicine (including acute respiratory illnesses), possibly due to increased Reactive Oxygen Species (ROS) production: ROS can cause oxidative stress and damage proteins, DNA, and lipids. Observational data from our group shows most surgical patients currently receive nearer 55% O2 under GA. The effect of intraoperative O2 concentration on other surgical outcomes remains unknown.

This project will determine whether giving lower concentrations of oxygen to surgical patients during anaesthesia can reduce levels of oxidative stress during surgery (particularly in the lungs); investigate how this affects other organs; and evaluate the feasibility of performing a large (multi-centre) effectiveness study to define 'safe' oxygen administration concentrations during surgery.

Patient undergoing elective major surgery will be randomised to receive 80% (WHO's recommendation); 55% (current usual care) or 30% oxygen (intervention) throughout anaesthesia. Endotracheal aspirates will be sampled along with paired central venous and arterial blood samples throughout surgery to monitor levels of oxidative stress and organ function. Patients will be followed up for 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16yrs - no upper limit
* Undergoing elective surgical procedure
* Planned for placement of arterial line and central venous catheter as part of routine anaesthetic delivery
* Written informed consent

Exclusion Criteria:

* Withdrawal of written consent or unable to give informed written consent
* Pregnant at time of enrolment
* Neurosurgery, cardiothoracic surgery or any other operation involving 1 lung ventilation at any point during procedure
* Baseline SpO2 < 90%
* Severe COPD (3 or 4 on GOLD criteria), Interstitial lung disease or other severe respiratory inflammatory co-morbidity (including already on home oxygen)
* BMI > 35
* Assessed as having a potentially difficult airway or being difficult to ventilate (defined as concern documented at anaesthetic assessment)
* Participating in another research trial with similar interventions or outcomes.
* Sickle cell disease
* Thalassemia Major
* Under custody

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total Free Thiols | End of surgery
  A measure of (Anti)oxidant capacity

SECONDARY OUTCOMES:
Other oxidative stress markers | Within 7 days of surgery
  A panel of other markers of oxidative stress
Acute cardiac events | Within 7 days of surgery
  Elevations in troponin levels
Acute Kidney Injury | Within 7 days of surgery
  Elevations in creatinine or NGAL-1
Acute Liver Injury | Within 7 days of surgery
  Elevations in ALT
Post-operative Cognitive Recovery | 7 days after surgery
  PQRS score
Postoperative Morbidity | 7 days after surgery
  Post Operative Morbidity Survey score

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cumpstey, BM BCh, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided